CLINICAL TRIAL: NCT01440023
Title: Developing Effective Response Inhibition Training for Symptom Relief in Tourette Syndrome
Brief Title: Developing Cognitive Training for Tourette Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Collaborators: Tourette Association of America (Other)
Responsible Party: Principal Investigator, Han Joo Lee, Assistant Professor of Clinical Psychology, University of Wisconsin, Milwaukee
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TSA-2011-Lee; TSA (Other: Tourette Syndrome Association)
Record Dates: First submitted 2011-09-02; First posted 2011-09-23 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Tourette Syndrome; Chronic Tic Disorders
Keywords: tic disorder; tourette syndrome; habit reversal; response inhibition; cognitive retraining
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBIT + Response Inhibition Training (Experimental): CBIT is an 8 session treatment protocol held over 10 weeks. In CBIT, core components are implemented across the various therapy sessions. These core components include habit reversal training (HRT), functional assessment/function-based interventions, and a behavioral reward program for the child. Each core component is briefly described below. HRT/CBIT involves three components, awareness training, competing response training, and social support training (Woods, Twohig, Roloff, & Flessner, 2003). For this condition, CBIT will be combined with adjunctive computerized response inhibition training, which will be delivered over the first 4 weeks of the CBIT treatment.
  Interventions: Behavioral: Comprehensive Behavioral Intervention for Tics (CBIT); Behavioral: Computerized Response Inhibition Training
- Experimental: CBIT + Placebo Computer Training (Placebo Comparator): In this condition, participants receive the same package of CBIT treatment, which consists of awareness training, competing response training, and social support training (Woods, Twohig, Roloff, & Flessner, 2003). Additionally, the standard CBIT treatment is combined with computer-based placebo cognitive training that is irrelevant to the target cognitive ability (i.e., response inhibition). During the first 4 weeks of the CBIT treatment, participants will receive 8 sessions of placebo cognitive training.
  Interventions: Behavioral: Comprehensive Behavioral Intervention for Tics (CBIT); Behavioral: Computerized Placebo Cognitive Training

INTERVENTIONS:
Behavioral: Comprehensive Behavioral Intervention for Tics (CBIT) — CBIT is an 8 session treatment protocol held over 10 weeks. Its core components are implemented across the various therapy sessions. These core components include habit reversal training (HRT), functional assessment/function-based interventions, and a behavioral reward program for the child.
  Other Names: Habit Reversal for Tourette Syndrome
Behavioral: Computerized Response Inhibition Training — Twice-weekly 45 minute computerized sessions for cognitive training focused on enhancing response inhibition capabilities.
  Arms: CBIT + Response Inhibition Training
Behavioral: Computerized Placebo Cognitive Training — Twice-weekly 45 minute computerized sessions for placebo cognitive training, which has been designed to be irrelevant for response inhibition capabilities.
  Arms: Experimental: CBIT + Placebo Computer Training

SUMMARY:
Many researchers suspect that individuals with Tourette Syndrome (TS) may have a poor cognitive ability (i.e., response inhibition; RI) that is essential to inhibit inappropriate response such as vocal or motor tics. The investigators aim to test whether a well-established behavior therapy for TS can be improved by increasing the individual's RI capabilities. To this end, 20 children will be randomly assigned to behavior therapy with computer-based RI training or behavior therapy with placebo computer-based cognitive training. The investigators will test the hypothesis that computer-based RI training can be a useful addition to the well-established behavior therapy to enhance its therapeutic effect.

DETAILED DESCRIPTION:
The current research seeks to examine the feasibility of using a computer-based RI training program as an adjunctive intervention for the Comprehensive Behavioral Intervention for Tics (CBIT). Our central hypothesis is that cognitive training designed to enhance RI will potentiate treatment outcomes of CBIT. To this end, the investigators will conduct a two-arm placebo-controlled double-blind trial, in which 20 children with TS will be randomly assigned to CBIT with computerized RI training (CBIT+RIT; n=10) or CBIT with placebo computer training (CBIT +PLT; n=10). CBIT consists of eight weekly sessions that present awareness training, competing response training, relaxation training and functional contingency management in a manualized format. The adjunctive computer training (RIT or PLT) will be delivered during the first 4 weeks of CBIT/HRT (i.e. 8 twice-weekly 40-min sessions). Tic symptoms and RI capabilities will be assessed at baseline, mid-treatment, post-treatment, and 1 month follow-up. This project is expected to increase our understanding about the nature of response inhibition deficits in TS and generate knowledge that will guide the development of effective cognitive interventions for TS.

ELIGIBILITY:
Inclusion Criteria:

* age between 9 and 17
* a diagnosis of TS or chronic tic disorder on the structured diagnostic interview
* moderate to severe levels of tic symptoms (YGTSS total score > 13 for TS, or > 9 for CTD), and (d) IQ > 80.

Exclusion Criteria:

* current substance abuse or dependence
* current or past psychotic disorder, bipolar disorder, or schizophrenia
* 4 or more previous sessions of behavioral treatments for tic
* significant suicidal ideation and/or attempts within the past 3 months
* any recent (in the previous month) or planned change in medication for tic symptoms.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in scores on the Yale Global Tic Severity Scale (YGTSS) across baseline, 4-week, 8-week, and 12 week assessments. during and after the treatment from baseline | At baseline, 4 week (mid-treatment), 8 week (post-treatment), and 12 week (1-month follow-up)
  The YGTSS is a well-validated instrument that produces severity ratings for motor and vocal tics, impairment caused by the tics, and an overall severity score of tic symptoms.

SECONDARY OUTCOMES:
Change in scores on the Clinical Global Impression Severity and Improvement (CGI-S and CGI-I) across baseline, 4-week, 8-week, and 12 week assessments. | At baseline, 4 week (mid-treatment), 8 week (post-treatment), and 12 week (1-month follow-up)
  The CGI-S and CGI-I are clinicianadministered rating scales that have been widely used in treatment outcome research for over 25 years. The current research will use the CGI scale to evaluate the overall severity and improvement in tic symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Han Joo Lee, Ph.D., Principal Investigator — University of Wisconsin, Milwaukee
Locations (1):
- The Psychology Clinic, University of Wisconsin-Milwaukee, Milwaukee, Wisconsin, United States